CLINICAL TRIAL: NCT07021833
Title: Multicenter Pilot Study of the Cryosa System for the Treatment of Obstructive Sleep Apnea (ARCTIC_AUS)
Brief Title: Clinical Trial of the Cryosa System for the Treatment of Obstructive Sleep Apnea (ARCTIC_AUS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cryosa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12458
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cryosa Procedure (Experimental)
  Interventions: Device: Cryosa Procedure

INTERVENTIONS:
Device: Cryosa Procedure — The purpose of this study is to evaluate the safety and effectiveness of Cryosa System applied to the tongue and soft palate in patients with clinically diagnosed obstructive sleep apnea (OSA).

SUMMARY:
This is a prospective, multicenter, non-randomized single-arm safety and performance study to collect data to evaluate the safety of the Cryosa procedure to treat obstructive sleep apnea (OSA) in patients with moderate to severe OSA. The study will also evaluate the chronic performance of the Cryosa system and collect clinical measures for therapy effectiveness that will be used to demonstrate safety and effectiveness in the next clinical study.

DETAILED DESCRIPTION:
The study will treat up to 30 subjects at up to 5 sites in Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of providing informed consent
2. Willing and capable of receiving the study procedure and returning for all follow-up evaluations and sleep studies
3. Willing and capable of completing all questionnaires
4. Age is 22 to 70 years old
5. Not able to use, refuse to use, or intolerant of Positive Airway Pressure (PAP) or Mandibular Advancement Devices (MAD)
6. BMI of ≤ 40 kg/m2 at enrollment
7. AHI >=30 at enrollment based on in-lab polysomnography study OR AHI ≥ 15 and BMI of >= 30 at enrollment based on in-lab polysomnography study

Exclusion Criteria:

General Exclusions

1. Subject currently participating in other premarket investigational studies unless approved by Sponsor in writing
2. Any reason the investigator deems the subject unfit for participation in the study

   Concomitant Medication Exclusions
3. Actively taking ACEs/ARBs for hypertension AND is either of black race, of female gender or >65 years of age
4. Actively undergoing immunotherapy (Allergy shots), or unwilling to washout of allergy shots at least 2 weeks prior to study procedure
5. Patients taking any of the following medication that could affect study endpoints: benzodiazepines, Z-drugs (zolpidem and eszopiclone) opiates, antipsychotics (neuroleptics), phenothiazines, and prescription stimulants (including Sunosi, Provigil, and Nuvigil)
6. Currently on stable GLP-1 medication dosing and unwilling to commit to maintaining that dose until completion of the 6-month assessment post-procedure.
7. Currently titrating GLP-1 medication and unwilling to discontinue use 1 month prior to procedure date and commit to not to re-start until completion of the 6-month assessment post-procedure

   Medical History Exclusions
8. Prior sleep surgeries, including tongue base reduction or palatoplasty (with exception of tonsillectomy and/or adenoidectomy)
9. Previous surgery (non-OSA) within 12 weeks of scheduled procedure performed on the soft tissue of the upper airway (e.g., uvula, soft palate, or tonsils)
10. Patients with severe, uncontrolled asthma
11. History of angioedema/swelling of the airway
12. Hereditary angioedema and other autoimmune disorders that could lead to acquired angioedema confirmed with a compliment component C4 blood test <13mg/dL
13. History or presence of cold urticaria at the time of screening
14. History of cryoglobulinemia
15. History of allergy to glycerin
16. Diagnosed autoimmune disorders including active thyroid disease, lupus, multiple myeloma, chronic lymphocytic leukemia
17. Oral cancer or non-healing oral wounds
18. History of radiation therapy to neck or upper respiratory tract
19. Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat (with exception of tonsillectomy and/or adenoidectomy)
20. Resistant hypertension, defined as a blood pressure that remains above goal despite concurrent use of three antihypertensive agents of different classes taken at maximally tolerated doses
21. Neuromuscular disease or other neurologic deficits (for example multiple sclerosis, muscular dystrophy, Parkinson's disease, transient ischemic attack, epilepsy or cerebrovascular accident)
22. Diagnosis of any moderate to severe congestive obstructive pulmonary disease (COPD)
23. Active, severe pulmonary vascular disease (for example pulmonary arterial hypertension or pulmonary embolism)
24. Uncontrolled Diabetes (including Diabetes Mellitus [DM] or Insulin Dependent Diabetes Mellitus [IDDM]) with HbA1c >9
25. Currently receiving treatment for severe cardiac valvular dysfunction, NYHA Class III or IV heart failure, unstable angina or recent (< 12 months) myocardial infarction or severe cardiac arrhythmias
26. Subjects with bleeding event, known bleeding diathesis, impaired immunity for any reason, or heart attack or stroke within the last 12 months
27. Clinical evidence of severe renal failure (Stage 4 or 5) undergoing dialysis or expected to institute dialysis within 6 months
28. History or current clinical evidence of TIA or stroke or muscular dysfunction
29. Other severe sleep disorders that in the opinion of the investigator, confound functional assessments of sleepiness such as narcolepsy with cataplexy, severe insomnia/insomnia secondary to chronic pain, PTSD
30. Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject's ability to meet study requirements and ability to provide study consent

    Lifestyle / Work
31. Current smoker (≥ 1 pack/day)
32. Presence of occupational shift work or anticipation of shift changes during the study duration
33. Subject has sleep hygiene behavior that is likely to interfere with measurement outcomes during PSG.
34. Known active substance use disorder
35. Females who are pregnant or females of childbearing age with intention to become pregnant during the study period (period defined as ≤ 3 months from treatment date)
36. Unwilling or unable to refrain from and washout use of oral appliances or positional devices for the PSG sleep studies.
37. Unwilling or unable to refrain from use of PAP, oral appliances for OSA, OSA surgery, or medications for OSA from enrollment through the completion of the Month 6 follow-up visit
38. Subject has an occupation for which untreated OSA presents a substantial risk to safety
39. Residing at or is planning to move within 2 years to a location where the subject would no longer be willing or capable of returning for all follow-up evaluations and sleep studies.

    Upper Airway Exam
40. Severe maxillary mandibular insufficiency that in the opinion of the investigator thought to be the primary cause of OSA
41. Obvious severe fixed upper airway obstructions (tumors, polyps, nasal obstruction)
42. Obstructions identified at the tonsils (palatine tonsils size 3+ or 4+)
43. Lingual tonsils size 4+
44. Friedman tongue position IV

    Surgical Consult
45. Contraindication to general anesthesia or in the opinion of the Investigator would not be able to tolerate the procedure, including intubation during the procedure
46. Any reason for which, in the judgment of the investigator, the subject is considered to be a poor surgical or study candidate, which may include, but is not limited to: any medical, anatomical, social, or psychological problems that could complicate the procedure and/or recovery from the procedure or could complicate the required procedures and evaluations of the study

    PSG Exclusion Criteria
47. ≥ 25% Central and mixed apnea and hypopnea events as a proportion of the sum of apnea and hypopnea events per hour
48. Oxygen saturation must be ≥ 70% for ≥ 90% of time during sleep.
49. Non-supine AHI < 10, minimum of 45 minutes non-supine sleep time
50. Failure to complete a 72-hour CPAP washout period before administering the PSG and unwilling to repeat

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Procedure or Device/Treatment Related Events | 90 days post procedure
  Safety will be assessed by evaluating all serious procedure- or device/treatment-related events occurring in the first 90 days post-procedure

IPD SHARING:
Plan to Share IPD: No